CLINICAL TRIAL: NCT05445206
Title: Clinical Validation Study for Noninvasive Cardiopulmonary Management Device (Phase II)
Brief Title: Clinical Validation Study for CPM Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Analog Device, Inc. (Other)
Collaborators: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Resp CPM Validation
Record Dates: First submitted 2022-06-30; First posted 2022-07-06 (Actual); Results first posted 2024-06-12 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: Comparison between test device and reference device
Masking Description: The individuals who annotate the capnography waveform are blinded between the reference strip and the test device strip.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Health Adult (Experimental): The target population is healthy adult volunteers who do not have preexisting heart or lung conditions or illness. The goal is to recruit a participant population with a range of body types and BMIs and an approximately even split of genders.
  Interventions: Device: CardioPulmonary Management Device (CPM)

INTERVENTIONS:
Device: CardioPulmonary Management Device (CPM) — CPM device is used in tangent with reference capnography device.

SUMMARY:
This study is designed to be a clinical validation study to ready the CPM System for FDA 510(k) submission. This study will be conducted as a prospective non-randomized. The study is non-significant risk since the CPM Device is noninterventional and noninvasive. The study is primarily designed to validate the accuracy of the respiration rate and the changes in relative tidal volume. All participants will be fitted with both the CPM Device as well as reference devices (capnography and ECG). Participants will be randomized between 4 procedures (A-D) which will determine the order of 18 exercises. Each exercise has about 2 minutes of device recording and two minutes of rest. Each exercise contains two positions: sitting up for one minute and lying down for one minute. For some exercises, the participant will be instructed to breathe at a certain rate (assisted by a metronome). For other exercises, the participants will breathe at a normal rate but change how deep the are breathing. For exercise 18, all capnography reference devices will be removed, and an ECG reference device will be placed. After exercise 18, the participant will have all devices removed and the study visit will terminate. The participant will receive a safety follow-up call about 1 week after their visit.

ELIGIBILITY:
Inclusion Criteria:

* Adults over the age of 18 and who are willing and able to give informed consent
* Willing and able to participate in all activities related to this study, including trimming chest hair and wearing a reference device and the CPM wearable device
* Volunteers of any race, any gender
* Range of physiques
* Healthy

Exclusion Criteria:

* Injury or skin disturbance in the area of the test device
* Allergies or sensitivities to silicone/acrylic-based adhesive
* Pregnant, method of assessment at discretion of PI
* Currently smokes cigarettes
* Has known respiratory conditions that might prevent them from following the study procedure such as:

  * Flu
  * Pneumonia/bronchitis
  * Shortness of breath/respiratory distress
  * Respiratory or lung surgery
  * Emphysema, COPD, lung disease
* Has self-reported heart or cardiovascular conditions such as chest pain, AFib, CHF, cardiomyopathy, or other conditions that could interfere with cardiopulmonary function
* Has other self-reported health conditions that could interfere with the breathing patterns and exercises detailed in the protocol (including wearing a capnography mask)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-03-02 (Actual); Primary Completion 2022-07-06 (Actual); Study Completion 2022-07-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic Hospital, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Health Adult
Started | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Health Adult
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.2 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 39
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 36
  More than one race | 0
  Unknown or Not Reported | 0
BMI [Mean (Standard Deviation); unit: kg/m^2] | 26.7 (6.0)
Height [Mean (Standard Deviation); unit: centimeters] | 171.4 (10.3)
Weight [Mean (Standard Deviation); unit: kilograms] | 78.2 (17.9)

OUTCOME MEASURES:

1. Primary Outcome: Accuracy of CPM System Calculated RR Versus Reference Device Via Percent of Error Accuracy of Respiration Rate
Description: Accuracy of CPM System calculated RR versus reference device reported as percentage of respiration rate error within +/- breath rates per minute. Acceptance for clinical utility is >= 85%. Percentage of respiration rate error within ± 2bpm. Acceptance criteria for clinical utility is >= 85%. The percentage of respiration rate within ± 2brpm was calculated by data points, regardless of its rate and breathing condition, which the CPM System did not screen, therefore reporting the numeric values. Each data point will produce binary result (True or False) if the error is within ± 2 brpm. Assuming this binary result follows a binominal distribution, its confidence interval is also calculated.
Time Frame: up to 3 hours
Measure: Number (95% Confidence Interval); unit: Percent
Units Other Than Participants: device measurements
Groups:
- Supine Position Measurements: This arm includes measurements taken in position 1 of a CPM system device reading (supine position).
- Upright Position Measurements: This arm includes measurements taken in position 2 of a CPM system device reading (upright position).
Arm/Group | Supine Position Measurements | Upright Position Measurements
Number analyzed (Participants) | 40 | 40
Number analyzed (device measurements) | 716 | 716
Percent | 96.3 [94.5 to 97.6] | 95.7 [93.8 to 97.2]

2. Primary Outcome: Root Mean Squared Error (RMSE) of Respiration Rates From the CPM System vs Reference Device for Metronome Guided Breathing and Non-metronome Guided Breathing.
Description: Root mean square (RMS) of residual relative error of relative tidal volume. Acceptance criteria for clinical utility is <= 35%. First, the subject-specific linear fitting is performed after taking the natural log of both CPM's rTV and reference TV. Then, the residual errors in rTV after the fitting were calculated. Finally, all subject's residual errors are pooled together to calculate the root mean squared (RMS) residual relative errors. The confidence interval was calculated assuming the square of this error follows Chi-square distribution. This error characterized in a log-log domain is converted back to characterize a relative accuracy by taking an exponential of natural constant followed by subtraction of one. The RMS of residual error in % is characterized in this way because the linear fitting in the log-log domain and its residual errors represents faithful relative residual error regardless of an absolute value of TV.
Time Frame: up to 3 hours
Measure: Number (95% Confidence Interval); unit: Percent RMS residual relative error
Units Other Than Participants: device measurements
Arm/Group | Supine Position Measurements | Upright Position Measurements
Number analyzed (Participants) | 40 | 40
Number analyzed (device measurements) | 716 | 716
Percent RMS residual relative error | 23.6 [22.2 to 25.3] | 32.6 [30.4 to 35.0]

3. Secondary Outcome: Accuracy of CPM System Calculated Respiration Rate Versus Reference Device, Reported as Root Mean Squared (RMS) Error
Description: Accuracy of CPM System calculated RR versus reference device. It is reported in Root Mean Squared error for both exercises with metronome guided breathing and non-metronome guided breathing. Acceptance criteria of substantial equivalence is ~1.6 breath rates per minute (BRPM) for metronome guided breathing and 3.0 BRPM for non-metronome guided breathing.
Time Frame: up to 3 hours
Measure: Number; unit: BRPM
Units Other Than Participants: relative tidal volume data points
Arm/Group | Supine Position Measurements | Upright Position Measurements
Number analyzed (Participants) | 36 | 36
Number analyzed (relative tidal volume data points) | 570 | 546
BRPM
  Root Mean Squared Error - Metronome Guided breathing | 1.09 | 1.29
  Root Mean Squared Error - Non-Metronome Guided breathing | 0.91 | 1.91

4. Secondary Outcome: CPM's ECG Metrics Compared to Reference Device Lead II ECG Metrics (Results Displayed as % Comparasion)
Description: Test the CPM System ECG strip against a lead II ECG strip. Results are displayed as % of CPM strips equivalent to Lead II ECG strips. One CPM ECG strip and one reference lead II strip were analyzed per patient.
Time Frame: up to 3 hours
Population: Subject's ECG strips that did not pass the quality check were not included in the analysis, leading to a different number of participants than for the respiration parameters.
Measure: Number; unit: Percent
Units Other Than Participants: strips analyzed
Arm/Group | Health Adult
Number analyzed (Participants) | 29
Number analyzed (strips analyzed) | 58
Percent
  Quality QRS presentation | 100
  QRS width measurability | 100
  Accurate Determination of QRS widening | 94.9
  QT interval measurability | 100
  A-Fib Rhythm readability | 100

5. Secondary Outcome: Test Device Skin Temperature vs Reference Device Skin Temperature Comparison
Description: The accuracy is characterized as mean error across all measurement items and all subjects.
Time Frame: up to 3 hours
Measure: Mean (Standard Error); unit: degrees Celcius
Arm/Group | Health Adult
Number analyzed (Participants) | 40
degrees Celcius | 0.02 (.81)

ADVERSE EVENTS:
Time Frame: 1 week
Arm/Group | Health Adult
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-02-07): https://cdn.clinicaltrials.gov/large-docs/06/NCT05445206/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-12): https://cdn.clinicaltrials.gov/large-docs/06/NCT05445206/SAP_002.pdf